CLINICAL TRIAL: NCT02504099
Title: Open-label Study to Evaluate the Safety and Efficacy of the Combination of Ombitasvir, Paritaprevir/r ± Dasabuvir With or Without Ribavirin (RBV) in Adult Patients With GT1 or GT4 Chronic HCV Infection and Response to Prior Treatment of Early Stage Hepatocellular Carcinoma (GEODE - I)
Brief Title: A Study to Evaluate the Safety and Efficacy of Ombitasvir/Paritaprevir/r With or Without Dasabuvir and With or Without Ribavirin in Chronic Hepatitis C Virus Genotype 1 or 4 Infected Adults With Successfully Treated Early Stage Hepatocellular Carcinoma
Acronym: GEODE - I
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study stopped due to low enrollment
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M14-726; 2015-001049-10 (EudraCT Number)
Record Dates: First submitted 2015-07-20; First posted 2015-07-21 (Estimated); Results first posted 2017-12-12 (Actual); Last update posted 2017-12-12 (Actual); Status verified 2017-11

CONDITIONS: Chronic Hepatitis C Infection
Keywords: Chronic Hepatitis C Infection; Early Stage Hepatocellular Carcinoma
MeSH Terms: interventions — ombitasvir; dasabuvir; Viekira Pak; paritaprevir; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- OBV/PTV/r ± DSV ± RBV for 12 or 24 weeks (Experimental): OBV/PTV/r (ombitasvir/paritaprevir/ritonavir [25 mg/150 mg/100 mg once daily]) with or without dasabuvir (250 mg twice daily) with or without weight-based ribavirin (± RBV; dosed 1,000 or 1,200 mg daily divided twice a day) for 12 or 24 weeks, dosed as per label based on HCV genotype/subtype and presence of cirrhosis.
  Interventions: Drug: ombitasvir/paritaprevir/ritonavir and dasabuvir; Drug: ombitasvir/paritaprevir/ritonavir; Drug: ribavirin

INTERVENTIONS:
Drug: ombitasvir/paritaprevir/ritonavir and dasabuvir — Tablet; ombitasvir coformulated with paritaprevir and ritonavir, dasabuvir tablet
  Other Names: Viekira Pak; paritaprevir also known as ABT-450; ombitasvir also known as ABT-267; dasabuvir also known as ABT-333
Drug: ombitasvir/paritaprevir/ritonavir — Tablet; ombitasvir coformulated with paritaprevir and ritonavir
  Other Names: Technivie; paritaprevir also known as ABT-450; ombitasvir also known as ABT-267
Drug: ribavirin — Tablet

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of ombitasvir/paritaprevir/ritonavir (OBV/PTV/r), with or without dasabuvir (DSV) coadministered with or without ribavirin (RBV) for 12 or 24 weeks in adult patients with genotype 1 or genotype 4 chronic HCV infection and treated early stage Hepatocellular Carcinoma with compensated cirrhosis.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, at least 18 years of age at time of screening
2. Chronic hepatitis C virus (HCV) infection prior to study enrollment with screening laboratory results indicating HCV genotype 1 or 4 infection
3. Early stage hepatocellular carcinoma (HCC) diagnosed based on the typical hallmark of HCC (hypervascular in the arterial phase with washout in the portal venous or delayed phases)
4. Compensated cirrhosis defined as a Child-Pugh score of 5 or 6 at Screening

   • A minimal rim of ascites if detected at imaging is acceptable. Exclude ascites that requires the need to apply diuretic treatment to control ascites
5. Documented complete response to HCC treatment.
6. Females must be post-menopausal for more than 2 years or surgically sterile or practicing acceptable forms of birth control.

Exclusion Criteria:

1. Use of known strong or moderate inducers of cytochrome P450 3A (CYP3A) in participants receiving ombitasvir/paritaprevir/ritonavir (OBV/PTV/r) with and without dasabuvir (DSV), strong inducers and inhibitors (e.g., gemfibrozil) of cytochrome P450 2C8 (CYP2C8) in participants receiving OBV/PTV/r with DSV, medications contraindicated for ritonavir or RBV (for those that receive RBV) within 2 weeks or 10 half-lives (if known), whichever is longer, prior to study drug . For medications contraindicated with AbbVie's 2-direct-acting antiviral agent (2-DAA) and 3-DAA regimen, refer to the recommended prescribing information section of the approved local product labels.
2. Positive test result for hepatitis B surface antigen (HBsAg) or anti-human immunodeficiency virus antibody (HIV Ab).
3. Patients regardless of eligibility to liver transplant, who have a comorbid disease that might preclude completion of study follow-up.
4. Clinically significant abnormalities, other than HCV infection, in a participant with HCC based upon the medical history, physical examination, vital signs, laboratory profile and a 12-lead electrocardiogram (ECG) that make the participant an unsuitable candidate for this study in the opinion of the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2015-07; Primary Completion 2016-09 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc, Study Director — AbbVie

REFERENCES:
- See also: Related Info — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | OBV/PTV/r ± DSV ± RBV for 12 or 24 Weeks
Started | 3
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | OBV/PTV/r ± DSV ± RBV for 12 or 24 Weeks
Number analyzed (Participants) | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.3 (1.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Virologic Response 12 Weeks Post-treatment (SVR12)
Description: SVR12 was defined as plasma hepatitis C virus ribonucleic acid (HCV RNA) level less than the lower limit of quantification [<LLOQ]) 12 weeks after the last dose of study drug. Participants with missing data after flanking imputation were imputed as nonresponders.
Time Frame: 12 weeks after the last actual dose of study drug
Population: The data collected were not sufficient to analyze primary or secondary outcome measures. Only safety data were reported.
Arm/Group | OBV/PTV/r ± DSV ± RBV for 12 or 24 Weeks
Number analyzed (Participants) | 0

2. Secondary Outcome: Percentage of Participants With On-treatment Virologic Failure
Description: On-treatment virologic failure was defined as confirmed HCV RNA ≥ LLOQ after HCV RNA < LLOQ during treatment; confirmed increase of > 1 log(subscript)10(subscript) IU/mL above the lowest value post-baseline in HCV RNA during treatment; or HCV RNA ≥ LLOQ throughout treatment with at least 6 weeks of treatment.
Time Frame: Baseline (Day 1) and Treatment Weeks 2, 4, 8, 12 (end of treatment for 12-week treatment), 16, 20 and 24 (end of treatment for 12-week treatment)
Population: The data collected were not sufficient to analyze primary or secondary outcome measures. Only safety data were reported.
Arm/Group | OBV/PTV/r ± DSV ± RBV for 12 or 24 Weeks
Number analyzed (Participants) | 0

3. Secondary Outcome: Percentage of Participants With Post-treatment Relapse
Description: Post-treatment relapse was defined as confirmed HCV RNA ≥ LLOQ between the end of treatment and 12 weeks after the last dose of study drug among participants who completed treatment with HCV RNA levels < LLOQ at the end of treatment.
Time Frame: From the end of treatment through 12 weeks after the last dose of study drug
Population: The data collected were not sufficient to analyze primary or secondary outcome measures. Only safety data were reported.
Arm/Group | OBV/PTV/r ± DSV ± RBV for 12 or 24 Weeks
Number analyzed (Participants) | 0

4. Secondary Outcome: Percentage of Participants With Long Term Clinical Outcomes
Description: The percentage of participants with long term clinical outcomes (de novo hepatocellular carcinoma (HCC) lesions, liver decompensation, unexpected liver transplant, liver related death, or any of the above) from first dose of study drug through 24 weeks post-treatment follow-up.
Time Frame: up to 48 weeks
Population: The data collected were not sufficient to analyze primary or secondary outcome measures. Only safety data were reported.
Arm/Group | OBV/PTV/r ± DSV ± RBV for 12 or 24 Weeks
Number analyzed (Participants) | 0

5. Secondary Outcome: Percentage of Participants With Recurrent HCV Infection Post Liver Transplant
Description: The percentage of participants with recurrent HCV infection post liver transplant out of all participants with liver transplant during the study.
Time Frame: from liver transplant to 24 weeks post-treatment (up to 48 weeks)
Population: The data collected were not sufficient to analyze primary or secondary outcome measures. Only safety data were reported.
Arm/Group | OBV/PTV/r ± DSV ± RBV for 12 or 24 Weeks
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (TEAEs) and serious adverse events (TESAEs) were collected from first dose of study drug until 30 days after the last dose of study drug (up to 16 weeks for participants treated for 12 weeks and up to 28 weeks for participants treated for 24 weeks).
Description: TEAEs and TESAEs are defined as any adverse event that begins or worsens in severity after initiation of study drug until 30 days after the last dose of study drug.
Arm/Group | OBV/PTV/r ± DSV ± RBV for 12 or 24 Weeks
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 3/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | OBV/PTV/r ± DSV ± RBV for 12 or 24 Weeks (N=3)
LEUKOPENIA (Blood and lymphatic system disorders) | 1
LYMPHOPENIA (Blood and lymphatic system disorders) | 1
NEUTROPENIA (Blood and lymphatic system disorders) | 1
DIARRHOEA (Gastrointestinal disorders) | 2
DYSPEPSIA (Gastrointestinal disorders) | 1
MESENTERIC VEIN THROMBOSIS (Gastrointestinal disorders) | 1
NAUSEA (Gastrointestinal disorders) | 1
PORTAL HYPERTENSIVE GASTROPATHY (Gastrointestinal disorders) | 1
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1
DEPRESSION (Psychiatric disorders) | 1
IRRITABILITY (Psychiatric disorders) | 1
NEPHROLITHIASIS (Renal and urinary disorders) | 1
PRURITUS (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.